CLINICAL TRIAL: NCT03465540
Title: A Phase 1 Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of AMG 397 in Subjects With Selected Relapsed or Refractory Hematological Malignancies
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of AMG 397 in Subjects With Selected Relapsed or Refractory Hematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decisions
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20170173
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma; Acute Myeloid Leukemia; Non-Hodgkins Lymphoma; Myelodysplastic Syndrome; AML; MDS; NHL
Keywords: Multiple Myeloma; Acute Myeloid Leukemia; Myelodysplastic Syndrome; AML; MDS; MM; Myeloid Cell Leukemia 1 Inhibitor; MCL1 Inhibitor; MCL1
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes | interventions — Dexamethasone; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1A: AMG 397 Dose Escalation (Experimental): This arm includes subjects with multiple myeloma (MM) or non-Hodgkin's lymphoma (NHL).
  Interventions: Drug: AMG 397
- Part 1B: AMG 397 Dose Escalation (Experimental): This arm includes subjects with acute myeloid leukemia (AML).
  Interventions: Drug: AMG 397
- Part 2A: AMG 397 Monotherapy (Experimental): This arm includes subjects with AML or myelodysplastic syndrome (MDS).
  Interventions: Drug: AMG 397
- Part 2B: AMG 397 Monotherapy (Experimental): This arm includes subjects with AML in Japan only.
  Interventions: Drug: AMG 397
- Part 2C: AMG 397 Monotherapy (Experimental): This arm includes subjects with MM.
  Interventions: Drug: AMG 397
- Part 3A: AMG 397 + Azacitidine Combotherapy (Experimental): This arm includes subjects MDS.
  Interventions: Drug: AMG 397; Drug: Azacitidine
- Part 3B: AMG 397+ Azacitidine Combotherapy (Experimental): This arm includes subjects AML.
  Interventions: Drug: AMG 397; Drug: Azacitidine
- Part 3C: AMG 397+ Dexamethasone Combotherapy (Experimental): This arm includes subjects MM.
  Interventions: Drug: AMG 397; Drug: Dexamethasone

INTERVENTIONS:
Drug: AMG 397 — AMG 397 will be administered orally once or twice weekly as part of a 28-day treatment cycle.
Drug: Dexamethasone — Dexamethasone will be administered intravenously (IV) or orally on Days 1, 8, 15, and 22 of each 28-day cycle.
  Arms: Part 3C: AMG 397+ Dexamethasone Combotherapy
Drug: Azacitidine — Azacitidine will be administered intravenously (IV) or subcutaneously (SC) daily for the first 7 days of a 28-day cycle.
  Arms: Part 3A: AMG 397 + Azacitidine Combotherapy; Part 3B: AMG 397+ Azacitidine Combotherapy

SUMMARY:
Evaluate the safety and tolerability of AMG 397. Estimate the maximum tolerated doses (MTDs) and/or biologically active doses.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), multicenter, non-randomized, open-label, phase 1 study evaluating AMG 397 administered orally once weekly, as part of a 28-day treatment cycle in adult subjects with selected relapsed or refractory hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Age ≥ 18 years old
* Pathologically-documented, definitively-diagnosed relapsed or refractory multiple myeloma (MM), myelodysplastic syndrome (MDS), or acute myeloid leukemia (AML) and is intolerant to, or considered ineligible for available therapies known to provide clinical benefit
* MM subjects only: Measurable disease per the International Myeloma Working Group (IMWG) response criteria (assessed within 21 days prior to enrollment), as indicated by one or more of the following: cytogenic risk factor: 1q21 amplification/gain, serum M-protein ≥ 0.5 g/dL, Urine M-protein ≥ 200 mg/24 hours. For Subjects who do not meet 1 of the 2 prior criteria: Serum Free Light Chain (sFLC) ≥ 10 mg/dL (≥ 100 mg/L) and an abnormal sFLC ratio (< 0.26 or > 1.65) as per the IMWG response criteria
* MM subjects only: Hematological function, as follows without transfusion or growth factor support within 2 weeks prior to study day 1: absolute neutrophil count ≥ 1.0 X 109/L, hemoglobin > 8 g/dL and platelet count ≥ 75 X 109/L
* AML subjects only: Pathologically confirmed diagnosis of AML as defined by the World Health Organisation (WHO) Classification, more than 5% blasts in bone marrow and persisting or recurring following one or more treatment courses
* MDS subjects only: pathologically confirmed diagnosis of MDS as defined by the WHO Classification, intermediate and high risk MDS and intolerant or refractory to HMA treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Life expectancy of > 3 months, based on the opinion of the investigator
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption.
* Hepatic function, as follows:

  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN)
  * total bilirubin (TBL) < 1.5 X ULN (except subjects with Gilbert's syndrome)
* Cardiac function, as follows:

  * Cardiac ejection fraction ≥ 50% and no evidence of pericardial effusion as determined by echocardiogram or multigated acquisition (MUGA) scan
  * no ECG findings representing a recent cardiac injury within 6 months before enrollment
* Renal function as follows:

  * Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/minute calculated using the formula of Cockcroft and Gault [(140 - Age) × Mass (kg) / (72 × serum creatinine mg/dL)]. Multiply result by 0.85 if female

Exclusion Criteria:

Disease Related

* Previously received an allogeneic stem cell transplant within 6 months of study day 1 OR having signs or symptoms of acute or chronic graft-versus-host disease
* Autologous stem cell transplant < 90 days before enrollment
* Candidates for stem cell transplant should have failed or are not considered eligible for either allogeneic and autologous transplant

Other Medical Conditions

* History of other malignancy except:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 2 years before enrollment and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductal carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ
* Myocardial infarction within 6 months before enrollment
* Symptomatic congestive heart failure (New York Heart Association > Class II)
* History of arterial thrombosis (eg, stroke or transient ischemic attack) in the past 6 months before enrollment
* Uncontrollable active infection requiring intravenous anti-infective treatments within 1 week before enrollment
* Known positive results for human immunodeficiency virus (HIV)
* Active hepatitis B and C based on the following results: Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic, hepatitis B or recent acute hepatitis B), Negative HBsAg and positive for hepatitis B core antibody: hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B. Positive Hepatitis C virus antibody (HCVAb): hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C
* Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 grade 1, or to levels dictated in the eligibility criteria with the exception of grade 2peripheral neuropathy, alopecia or toxicities from prior anti-tumor therapy that are considered irreversible (defined as having been present and stable for > 4 weeks prior to study day 1 may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and sponsor)
* Antitumor therapy (chemotherapy, antibody therapy, molecular-targeted therapy, retinoid therapy, or investigational agent or procedures) within 14 days of day 1
* Prior systemic radiation therapy must have been completed at least 28 days before study day 1. Prior focal radiotherapy completed at 14 days before study day 1
* Females of reproductive potential who are unwilling to practice acceptable methods of highly effective contraception while on study through 8 months after receiving the last dose of study drug. Males who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use a condom with or without spermicide while on study through 5 months after receiving the last dose of study drug if sexually active with a female of childbearing potential
* Females who are lactating/breastfeeding or who plan to breastfeed while on study through 8 months after receiving the last dose of study drug
* Females with a positive pregnancy test or planning to become pregnant while on study through 8 months after receiving the last dose of study drug
* Males who are unwilling to abstain from sperm donation while on study through 8 months after receiving the last dose of study drug
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Use of any over-the-counter or prescription medications within 14 days or 5 half-lives (whichever is longer), prior to study day 1 that was not reviewed and approved by the principal investigator and the Amgen medical monitor
* Use of herbal medicines (eg, St. John's wort), vitamins, and supplements consumed by the subject within 14 days prior to study day 1 that was not reviewed and approved by the principal investigator and the Amgen medical monitor
* Use of any known inhibitors of P-gp within 14 days or 5 half-lives (whichever is longer) or grapefruit juice or grapefruit containing products within 7 days prior to study day 1 that was not reviewed and approved by the principal investigator and the Amgen medical monitor
* Use of known CYP3A4 sensitive substrates, (with a narrow therapeutic window), within 14 days or 5 half-lives (whichever is longer) of the drug or its major active metabolite, whichever is longer, prior to study day 1 that was not reviewed and approved by the principal investigator and the Amgen medical monitor
* Use of known P-gp substrates (with a narrow therapeutic window) within 14 days or 5 half-lives (whichever is longer) prior to study day 1 that was not reviewed and approved by the principal investigator and the Amgen medical monitor
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, long term follow-up) to the best of the subject and investigator's knowledge
* Known sensitivity to any of the products or component to be administered during dosing
* MM subjects with any of the following criteria are excluded:

  * Multiple myeloma with IgM subtype
  * POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
  * Existing plasma cell leukemia
  * Waldenstrom's macroglobulinemia
  * Amyloidosis
* AML subjects with the following criteria are excluded:

  * Circulating white blood cells > 25,000/μl. Hydroxyurea to control peripheral blood leukemic cell counts, within 24 hours of study day 1 is permitted
  * Promyelocytic leukemia
* AML/MDS subjects fit for intensive salvage therapy
* Subjects with elevated cardiac troponin above the manufacturer's 99th percentile upper reference limit for ADVIA Centaur XP assay at screening performed by the central laboratory (Covance)
* Subjects with evidence of recent cardiac injury at screening based on creatine kinase-muscle/brain (CK-MB), N-terminal prohormone of brain natriuretic peptide (NT-pro-BNP), and ECG assessments at screening
* Subjects with MDS that are eligible for hematopoietic stem cell transplant (HSCT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert and Med College Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- France (2):
  - Institut Paoli Calmettes, Marseille
  - Institut Gustave Roussy, Villejuif
- Alexandra Hospital, Athens, Greece
- Italy (2):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria di Bologna Policlinico S Orsola Malpighi, Bologna
- Ogaki Municipal Hospital, Ogaki-shi, Gifu, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 11 research centers in Australia, France, Greece and the United States from 17 August 2018 to 25 July 2019.
Pre-assignment Details: Parts 2 and 3 of the trial were not initiated after part 1 data was reviewed. No participants were screened or enrolled for parts 2 or 3.
Groups:
- Part 1a: 80 mg AMG 397: Participants with relapsed/refractory (RR) multiple myeloma (MM) and/or non-Hodgkin's lymphoma (NHL) received 80 mg AMG 397 once a day for 2 consecutive days followed by a 5 day break at a weekly interval (QD2), as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
- Part 1a: 160 mg AMG 397: Participants with RR MM and/or NHL received 160 mg AMG 397 QD2, as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
- Part 1a: 320 mg AMG 397: Participants with RR MM received 320 mg AMG 397 QD2, as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
- Part 1b: 80 mg AMG 397: Participants with RR acute myeloid leukemia (AML) received 80 mg AMG 397 QD2, as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
- Part 1b: 160 mg AMG 397: Participants with RR AML received 160 mg AMG 397 QD2, as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
- Part 1b: 320 mg AMG 397: Participants with RR AML received 320 mg AMG 397 QD2, as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
Period: Overall Study
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Started | 2 | 6 | 4 | 4 | 5 | 3
Received AMG 397 | 2 | 6 | 4 | 4 | 5 | 3
Completed (Completed Study) | 1 | 2 | 1 | 1 | 1 | 1
Not Completed | 1 | 4 | 3 | 3 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Death | 1 | 1 | 0 | 2 | 0 | 2
Not completed — Protocol specified criteria | 0 | 2 | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants who were enrolled and received at least 1 dose of AMG 397.
Groups:
- Part 1a: 80 mg AMG 397: Participants with RR MM and/or NHL received 80 mg AMG 397 QD2, as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
- Part 1b: 80 mg AMG 397: Participants with RR AML received 80 mg AMG 397 QD2, as part of a 28-day treatment cycle.
  Participants could receive AMG 397 until the participant became intolerant to the investigational product, signs and symptoms of clinical progression were evident as determined by the investigator, or the participant withdrew consent.
- Total: Total of all reporting groups
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397 | Total
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3 | 24
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 1 | 3 | 2 | 0 | 3 | 0 | 9
  From 65-84 years | 1 | 3 | 2 | 4 | 2 | 3 | 15
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 2 | 2 | 11
  Male | 1 | 4 | 3 | 1 | 3 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 6 | 3 | 4 | 4 | 3 | 22
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 5 | 3 | 4 | 3 | 1 | 18
  Other | 0 | 1 | 1 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: DLTs were defined as specific adverse events (AEs) that occurred in a participant during the DLT evaluation period (Day 1 to Day 28), that the investigator assessed as related to AMG 397. The grading and severity of AEs were based on the guidelines provided in the common terminology criteria for adverse events (CTCAE) version 4.03.
Time Frame: 28 days
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1.
  DLT evaluable set: All participants who experienced a DLT or who received at least 75% of the planned dose in the DLT window (Day 1 to Day 28).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 3 | 2
Participants | 0 | 0 | 1 | 0 | 0 | 1

2. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any AE starting on or after the first dose of investigational product. Any clinically significant changes in vital signs, physical examinations, electrocardiogram (ECGs) and clinical laboratory test results were recorded as AEs. The grading and severity of adverse events were based on the guidelines provided in the CTCAE version 4.03. Treatment-related TEAEs were any events that the investigator assessed as related to AMG 397.
Time Frame: Up to 30 days after last dose (Maximum time on treatment was 18 weeks for part 1a and 13 weeks for part 1b)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
Participants
  TEAEs | 2 | 6 | 4 | 4 | 5 | 3
  Treatment-related TEAEs | 2 | 6 | 4 | 2 | 4 | 3

3. Secondary Outcome: Overall Response Rate (ORR) for Participants With Multiple Myeloma (MM)
Description: ORR was assessed for participants with MM using response criteria per International Myeloma Working Group (IMWG).
  ORR was defined as the percentage of participants who experienced either one of the following based on investigator assessment:
  * partial response (PR)
  * very good partial response (VGPR)
  * complete response (CR)
  * stringent complete response (sCR)
Time Frame: Up to end of study (a maximum of 48 weeks)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1. Participants with MM were only enrolled in part 1a, so therefore data is only presented for part 1a.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397
Number analyzed (Participants) | 1 | 5 | 4
Percentage of participants | 0.0 [0.0 to 97.50] | 0.0 [0.0 to 52.18] | 0.0 [0.0 to 60.24]

4. Secondary Outcome: Overall Response Rate (ORR) for Participants With Non-Hodgkin's Lymphoma (NHL)
Description: ORR was assessed for participants with NHL using response criteria per Lugano Classification.
  ORR was defined as the percentage of participants who experienced either of the following based on investigator assessment:
  * partial metabolic response/ PR
  * complete metabolic response/ CR
Time Frame: Up to end of study (a maximum of 48 weeks)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1. Participants with NHL were only enrolled in part 1a, so therefore data is only presented for part 1a.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part 1a: Participants With NHL - 80 mg AMG 397: All participants in part 1a with NHL that received 80 mg AMG 397.
- Part 1a: Participants With NHL - 160 mg AMG 397: All participants in part 1a with NHL that received 160 mg AMG 397.
Arm/Group | Part 1a: Participants With NHL - 80 mg AMG 397 | Part 1a: Participants With NHL - 160 mg AMG 397
Number analyzed (Participants) | 1 | 1
Percentage of participants | 100.0 [2.50 to 100.00] | 0.0 [0.00 to 97.50]

5. Secondary Outcome: Overall Response Rate (ORR) for Participants With Acute Myeloid Leukemia (AML)
Description: ORR was assessed for participants with AML using response criteria per European Leukemia Network Response Criteria.
  ORR was defined as the percentage of participants who experienced either of the following based on investigator assessment:
  * PR
  * morphological leukemia-free state (MLFS)
  * complete remission with incomplete hematologic recovery (CRi)
  * complete remission
  * complete remission without minimal residual disease (CRmrd-).
Time Frame: Up to end of study (a maximum of 48 weeks)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1. Participants with AML were only enrolled in part 1b, so therefore data is only presented for part 1b.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 4 | 5 | 3
Percentage of participants | 0.0 (0.00) [0.00 to 60.24] | 0.0 (0.00) [0.00 to 52.18] | 0.0 (0.00) [0.00 to 70.76]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was calculated as time from first dose of investigational product date to disease progression date or death due to any cause, whichever was earlier.
  PFS time in months: (date of disease progression or death - first dose date +1)/30.4.
Time Frame: Up to end of study (a maximum of 48 weeks)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1. Per the statistical analysis plan (SAP), PFS was only to be calculated if the number of participants who experienced events (disease progression or death) was 10 or more in either part 1 or part 2.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
Months | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population.

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of investigational product date until death due to any cause.
  OS time in months: (date of death - first dose date +1)/30.4.
Time Frame: Up to end of study (a maximum of 48 weeks)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1. Per the SAP, OS was only to be calculated if the number of participants who experienced an event (death) was 10 or more in either part 1 or part 2.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
Months | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population.

8. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from the first dose of investigational product until the first documentation of objective response. Only participants who achieved an objective response were evaluated for TTR.
  TTR time in months: (date of the first observation of response - first dose of IP date +1)/30.4.
Time Frame: Up to end of study (a maximum of 48 weeks)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1. Per the SAP, TTR was only to be calculated if the number of participants who experienced an event (objective response) was 10 or more in either part 1 or part 2.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
Months | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population.

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR was only planned to be calculated for participants who achieved response (PR or better). DOR was defined as time from the first observation indicating a response to the subsequent date of disease progression or death, whichever was earlier.
  DOR time in months: (date of disease progression or death - date of the first observation of response +1)/30.4.
Time Frame: Up to end of study (a maximum of 48 weeks)
Population: Parts 2 and 3 were not initiated and did not enrol any participants, therefore results presented only included participants in part 1. Per the SAP, DOR was only to be calculated if the number of participants who experienced an event (objective response) was 10 or more in either part 1 or part 2.
  FAS: All participants who were enrolled and received at least 1 dose of AMG 397.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
Months | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population. | NA [NA to NA] — No data are available due to low event rate in the population.

10. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 397
Description: Predose data for Day 2 were analyzed/included with the Day 1 data.
Time Frame: Cycle 1 (cycle = 28 days): Predose, 1, 2, 3, 5, 8 & 12 hours postdose on Day 1; predose, 1, 2, 3, 5, 8, 12, 24 & 48 hours postdose on Day 2
Population: The Pharmacokinetic (PK) Analysis Set: All participants who received at least 1 dose of AMG 397 and had at least 1 PK sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
µg/mL
  Day 1 | 0.415 (0.470) [0.470 to 09.999] | 0.468 (0.606) [lower limit 0.606] | 0.908 (1.19) [lower limit 1.19] | 0.747 (0.785) [lower limit 0.785] | 1.31 (1.87) [lower limit 1.87] | 2.51 (2.83) [lower limit 2.83]
  Day 2 | 1.17 (1.29) [lower limit 1.29] | 1.80 (1.88) [lower limit 1.88] | 2.822 (3.17) [lower limit 3.17] | 1.41 (1.51) [lower limit 1.51] | 3.69 (4.46) [lower limit 4.46] | 4.57 (5.14) [lower limit 5.14]

11. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) for AMG 397
Description: Predose data for Day 2 were analyzed/included with the Day 1 data.
Time Frame: as for outcome 10
Population: The PK Analysis Set: All participants who received at least 1 dose of AMG 397 and had at least 1 PK sample collected.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
Hours
  Day 1 | 12 (12) [12 to 12] | 18 (8.0) [8.0 to 24] | 8.1 (5.1) [5.1 to 12] | 12 (8.1) [8.1 to 24] | 21 (7.8) [7.8 to 25] | 12 (11) [11 to 12]
  Day 2 | 4 (2.9) [2.9 to 5.1] | 8.3 (7.9) [7.9 to 12] | 7.9 (4.9) [4.9 to 8.2] | 6.6 (5.0) [5.0 to 8.1] | 7.2 (3.3) [3.3 to 8.5] | 8.1 (8.0) [8.0 to 12]

12. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to 168 Hours (AUC0-168) for AMG 397
Time Frame: Cycle 1 (cycle = 28 days): Predose, 3, 5, & 8 hours postdose on days 1 (12 hours postdose on Day 1 only), 8 & 15, predose & 8 hours postdose on Day 22 & days 2, 3, 4, 9, 16, 17, 18 & 23; Cycles 2, 3 & 4 (cycle = 28 days): Predose on days 2, 8, 15 & 22
Population: The PK Analysis Set: All participants who received at least 1 dose of AMG 397 and had at least 1 PK sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µg/mL
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
hr*µg/mL | 635 (70.8) [lower limit 70.8] | 115 (123) [lower limit 123] | 230 (266) [lower limit 266] | 108 (115) [lower limit 115] | 264 (306) [lower limit 306] | 227 (444) [lower limit 444]

13. Secondary Outcome: Clearance (CL) of AMG 397
Time Frame: as for outcome 12
Population: The PK Analysis Set: All participants who received at least 1 dose of AMG 397 and had at least 1 PK sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
L/hr | 1.08 (1.13) [lower limit 1.13] | 1.17 (1.21) [lower limit 1.21] | 1.02 (1.42) [lower limit 1.42] | 0.449 (0.488) [lower limit 0.488] | 0.563 (0.674) [lower limit 0.674] | 0.320 (0.467) [lower limit 0.467]

14. Secondary Outcome: Half-life (t1/2) of AMG 397
Time Frame: as for outcome 12
Population: The PK Analysis Set: All participants who received at least 1 dose of AMG 397 and had at least 1 PK sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 5 | 3
hours | 60.1 (62.8) [lower limit 62.8] | 49.7 (54.9) [lower limit 54.9] | 76.9 (90.1) [lower limit 90.1] | 96.3 (118) [lower limit 118] | 53.4 (55.1) [lower limit 55.1] | 109 (129) [lower limit 129]

ADVERSE EVENTS:
Time Frame: Mortality data are reported up to end of study (a maximum of 48 weeks); Adverse events are reported from Day 1 up to 30 days after last dose (Maximum time on treatment was 18 weeks for part 1a and 13 weeks for part 1b)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for the FAS.
Arm/Group | Part 1a: 80 mg AMG 397 | Part 1a: 160 mg AMG 397 | Part 1a: 320 mg AMG 397 | Part 1b: 80 mg AMG 397 | Part 1b: 160 mg AMG 397 | Part 1b: 320 mg AMG 397
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/6 | 0/4 | 2/4 | 0/5 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/2 | 4/6 | 2/4 | 4/4 | 4/5 | 3/3
Other Adverse Events (participants affected / at risk) | 2/2 | 6/6 | 4/4 | 4/4 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1a: 80 mg AMG 397 (N=2) | Part 1a: 160 mg AMG 397 (N=6) | Part 1a: 320 mg AMG 397 (N=4) | Part 1b: 80 mg AMG 397 (N=4) | Part 1b: 160 mg AMG 397 (N=5) | Part 1b: 320 mg AMG 397 (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1a: 80 mg AMG 397 (N=2) | Part 1a: 160 mg AMG 397 (N=6) | Part 1a: 320 mg AMG 397 (N=4) | Part 1b: 80 mg AMG 397 (N=4) | Part 1b: 160 mg AMG 397 (N=5) | Part 1b: 320 mg AMG 397 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 3 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 3 | 2 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 3 | 1 | 4 | 1
Oral blood blister (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Plicated tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3 | 1 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 2 | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Haemodilution (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 2 | 3 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT03465540/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03465540/SAP_001.pdf